CLINICAL TRIAL: NCT06227884
Title: Impact of Advanced Practical Nursing Intervention Versus Usual Care on Hypertension Control : Retrospective Single-center Quasi-experimental Study
Brief Title: Impact of Advanced Practical Nursing Intervention Versus Usual Care on Hypertension Control : Retrospective Study
Acronym: iIPArétro
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231667
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: Advanced practice nurse; Hypertension; Therapeutic adherence; Trial
MeSH Terms: conditions — Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with APN intervention: Participants with a schedule of a MD consultation (within approximately 2 to 12 months) + an APN intervention halfway between day hospitalization et MD consultation
  Interventions: Other: APN intervention
- Patients without APN intervention: Participants with a MD consultation only, within approximately 2 to 12 months
  Interventions: Other: No APN intervention

INTERVENTIONS:
Other: APN intervention — Participants with a schedule of a MD consultation (within approximately 2 to 12 months) + an APN intervention halfway between day hospitalization et MD consultation
  APN intervention is divided into five main steps:
  * clinical and paraclinical examinations,
  * appraisal of patient's knowledge,
  * health education on hypertension and treatments,
  * setting a written medication plan with the patient to invest him in his management with adjusting or renewing treatments identically if necessary
  * decision-making balance between the benefits and risks of non-adherence to medication. A time is scheduled at the end of the intervention to let the patient ask questions or express his difficulties if he needs to.
  Groups: Patients with APN intervention
Other: No APN intervention — Participants with a schedule of a MD consultation (within approximately 2 to 12 months)
  Groups: Patients without APN intervention

SUMMARY:
Hypertension is the most frequent chronic pathology in France and in the world. It is one of the main modifiable cardiovascular risk factors. In France, 50% of treated hypertensives are uncontrolled and only 30% of treated patients are fully adherent to their antihypertensive treatment. Poor adherence to drug treatments is considered as one of the main causes of non-control of hypertension.

Since 2018, a new profession has entered the French healthcare system: Advanced Practice Nurses (APN). They have many broad skills, at the interface of nursing and medical exercises.

The purpose of this interventional study is to assess the impact of APN on blood pressure (BP) control in the context of usual care of hypertension thanks to a better adhesion of patients and a better therapeutic alliance.

The hypothesis formulated is that an individual APN intervention, included in a usual hypertension management, improves BP control.

DETAILED DESCRIPTION:
Hypertension is the most frequent chronic pathology in France and in the world. It is one of the main modifiable cardiovascular risk factors. In France, 50% of treated hypertensives are uncontrolled and only 30% of treated patients are fully adherent to their antihypertensive treatment. Poor adherence to drug treatments is considered as one of the main causes of non-control of hypertension.

Since 2018, a new profession has entered the French healthcare system: Advanced Practice Nurses (APN). They have many broad skills, at the interface of nursing and medical exercises.

The purpose of this interventional study is to assess the impact of APN on blood pressure (BP) control in the context of usual care of hypertension thanks to a better adhesion of patients and a better therapeutic alliance.

The hypothesis formulated is that an individual APN intervention, included in a usual hypertension management, improves BP control.

This study will be a retrospective quasi-experimental study, conducted at the Diagnosis and Therapeutic Center of the Hôtel-Dieu University Hospital, Assistance Publique - Hôpitaux de Paris, France. The timeframe of the study should is from September 2020 to July 2023.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* being diagnosed with essential hypertension,
* being followed by a MD of the structure for hypertension management,
* having received a proposition to meet an APN for hypertension management between the day hospitalization and the next MD consultation,
* having received a loaned tensiometer with instructions during the day hospitalization and explanations for HBPM protocol.

Exclusion Criteria:

* being diagnosed with secondary hypertension,
* having APN follow-up before the day hospitalization,
* being lost to follow-up in the twelve months after the MD consultation
* not having the BP measurement by OBPM for the day hospitalization (baseline) and/or the endline (endline),
* pregnancy
* under guardianship or tutorship
* State Medical Help

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with essential hypertension, recruited in day hospitalization unit: HDJ CITE of the Hôtel-Dieu Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Blood pressure (BP) control | Between 2 to 12 months
  Blood pressure (BP) control in MD consultation
  * Rate of BP control (BP < 140/90 mmHg)
  * Mean (SD) of both systolic and diastolic BP

SECONDARY OUTCOMES:
Home blood pressure monitoring (HBPM) | Between 2 to 12 months
  Performance and quality of home BP monitoring (HBPM). 3-category variable: HBPM perfectly performed, HBPM poorly performed, and HBPM not performed.
Blood pressure (BP) control | Day hospitalization - Inclusion
  Evolution of BP control between day hospitalization and MD consultation. 3-category variable: now controlled, stable, no longer controlled
Blood pressure (BP) control | Between 2 to 12 months
  Evolution of BP control between day hospitalization and MD consultation. 3-category variable: now controlled, stable, no longer controlled
Therapeutic adjustments | Between 2 to 12 months
  Group with APN :
  Therapeutic adjustments and their indication(s) by the APN. Dichotomous variables: therapeutic adjustments (yes/no) and their indication(s): inefficacy (yes/no) and intolerance (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BLACHER, MD, PhD, Study Chair — Diagnosis and Therapeutic Center, Hôtel-Dieu University Hospital, Assistance Publique-Hôpitaux de Paris, Paris University, 75004 Paris
Locations (1):
- Diagnosis and Therapeutic Center, Hôtel-Dieu University Hospital, Assistance Publique-Hôpitaux de Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vay-Demouy J, Lelong H, Blacher J. Advanced Practice Nurse Intervention Versus Usual Care for Hypertension Control: A Pilot Open-Label Randomized Controlled Trial. J Clin Hypertens (Greenwich). 2025 May;27(5):e70068. doi: 10.1111/jch.70068. PMID 40346888